CLINICAL TRIAL: NCT03054103
Title: A Comparison of Midazolam vs. Midazolam/Ketamine for Conscious Sedation in Patients Undergoing Phacoemulsification Under Topical Anesthesia
Brief Title: Sedation Methods During Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00031444
Record Dates: First submitted 2017-02-02; First posted 2017-02-15 (Actual); Results first posted 2018-01-19 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Phacoemulsification; Cataract
Keywords: ketamine; midazolam; sedation
MeSH Terms: conditions — Cataract | interventions — Midazolam; Ketamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-masked, three-armed clinical comparison
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Surgical conditions and patient response not aware of medication given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Midazolam alone (Placebo Comparator): Drug: Midazolam titrated 0.5-2.0 mg + normal saline placebo. Midazolam + Normal saline
  Interventions: Drug: Midazolam + Normal saline
- Midazolam + Ketamine 5 mg (Active Comparator): Drug: Midazolam titrated 0.5-2.0 mg + Ketamine 10 MG/ML: 0.5 ML. Midazolam + Ketamine 10 MG/ML: 0.5 ML
  Interventions: Drug: Midazolam + Ketamine 10 MG/ML: 0.5 ML
- Midazolam + Ketamine 10 mg (Active Comparator): Drug: Midazolam titrated 0.5-2.0 mg + Ketamine 10 MG/ML: 1 ML. Midazolam + Ketamine 10 MG/ML: 1 ML
  Interventions: Drug: Midazolam + Ketamine 10 MG/ML: 1 ML

INTERVENTIONS:
Drug: Midazolam + Ketamine 10 MG/ML: 0.5 ML — 5 mg ketamine IV given just prior to onset of case. Then titrated midazolam up to 2 mg IV at beginning and during case.
  Other Names: Ketalar
  Arms: Midazolam + Ketamine 5 mg
Drug: Midazolam + Ketamine 10 MG/ML: 1 ML — 10 mg ketamine IV given just prior to onset of case. Then titrated midazolam up to 2 mg IV at beginning and during case.
  Other Names: Ketalar
  Arms: Midazolam + Ketamine 10 mg
Drug: Midazolam + Normal saline — Preoperative control: Normal saline placebo given preoperatively. Then protocol followed for titration of midazolam up to 2 mg IV at beginning and during case.
  Other Names: NS
  Arms: Midazolam alone

SUMMARY:
Background: Phacoemulsification is the most common surgical procedure performed in the United States and European Union and sedation is commonly used during phacoemulsification to help alleviate patient anxiety and prevent the patient from interfering with the procedure. The investigators have administered ketamine in addition to midazolam in this regard. To study the effectiveness of this technique, The investigators proposed a study to determine if adding low-dose ketamine to midazolam has any beneficial (or negative) effects on operating conditions, patient satisfaction, and recovery during and after unilateral phacoemulsification procedures performed using topical anesthesia and intravenous (IV) conscious sedation.

Methods: In a free-standing Outpatient Surgery Center, the investigators conducted a randomized, double-masked, 3-arm, prospective comparison of IV midazolam only vs. midazolam with ketamine 5 mg IV vs. midazolam with ketamine 10 mg IV. The investigators then measured a single surgeon's assessment of surgical conditions, self-reported patient satisfaction, postoperative pain score, and duration of postoperative stay. The investigators also analyzed the dose of midazolam required to meet subjective anxiolysis in each group.

DETAILED DESCRIPTION:
Phacoemulsification is the most common surgical procedure performed in the United States and European Union. In addition, the number of diagnoses of cataracts is expected to double from 25,000,000 in 2010 to 50,000,000 in 2050 while the incidence of phacoemulsification is also increasing. Therefore, any attempt to optimize outcome and efficiency is significant.

Sedation is commonly used during phacoemulsification to help alleviate patient anxiety and prevent the patient from interfering with the procedure. However, a great deal of variation exists in anesthetic management of these cases. Investigators have published use of a number of agents for sedation in the literature. These include midazolam, clonidine, propofol, fentanyl, dexmedetomidine, remifentanil, and oral diazepam. Intravenous (IV) clonidine has a half-life of 9-13 h and increased risk of postoperative hypotension. Propofol causes disinhibition and it has to be titrated during surgery to prevent oversedation. Opioids carry an increased risk of respiratory depression, prolonged sedation, as well as delirium in the elderly. Finally, oral medications do not allow for quick dose adjustments during surgery.

Intravenous midazolam is commonly used for sedation during phacoemulsification and other minor procedures. It has properties as an anxiolytic, muscle relaxant, and it is effective at reducing intraocular pressure. However, anxious patients administered benzodiazepines may require higher doses during cataract surgery which can lead to oversedation or disinhibition with subsequent patient movement. These responses can reduce the patient's ability to follow simple commands which can affect surgical outcome. Additionally, patients who receive too much sedation may fall asleep and wake up startled, similarly compromising the outcome of the surgery.

In the search for additional medications that can improve surgical conditions and patient comfort during phacoemulsification, the investigators explored the use of a medication that can improve analgesia and reduce patient movement during procedures, namely ketamine. Ketamine is an NMDA antagonist with both sedative and analgesic properties and has minimal effects on respiration. Ketamine has been used to premedicate and sedate patients undergoing day care procedures without adverse effects, and patients, typically, remain cooperative albeit being sedated. These properties along with its relatively short elimination half-life of 2 h (compared with 3-4 h for midazolam) make ketamine an attractive agent for sedation during monitored anesthesia care (MAC) for cataract surgery.

The purpose of this study was to determine if adding low-dose ketamine to midazolam has any beneficial (or negative) effects on operating conditions, patient satisfaction, and recovery during and after unilateral phacoemulsification procedures performed using topical anesthesia and IV conscious sedation.

The investigators measured the surgeon's assessment of the participant's cooperation during surgery according to a predetermined Likert scale. The investigators also recorded the following outcome measures regarding each participant's surgery: 1) total dose of midazolam, 2) average time spent in the procedural room, 3) postoperative length of stay (LOS), and 4) average postoperative pain score. The subjects received a survey inquiring about the subjects' comfort and sedation level during surgery. Finally, the investigators recorded the following demographic data for all participants: gender, age, psychiatric diagnoses, and use of CNS, psychiatric, or opioid medications.

Statistical Analysis The investigators used Fisher's exact test for examining data expressed as percentages, and Students t-test for yes/no data, and repeated measures ANOVA for 3 group analysis (LOS, surgical duration). The investigators judged significance at a P-value of 0.05. The investigators utilized a generalized estimated equations (GEE) to fit a logistic model to assess differences in the responses of patients based on amount of ketamine received. The GEE approach can fit models to correlated outcomes, as in the case where subjects had more than one procedure performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients met inclusion criteria if they were between 18- and 80-years-old and undergoing elective cataract surgery performed by a single ophthalmologist (KW).

Exclusion Criteria:

* Patients younger than 18, older than 80, those with a serum creatinine >3 mg/dl, advanced liver disease (liver enzymes twice the normal range or higher), and those with an allergy to any of the study medications were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2016-11-05 (Actual); Study Completion 2016-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy N Harwood, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Midazolam Alone: Drug: Titrated midazolam + normal saline placebo
  Normal saline: Preoperative control: Normal saline placebo given preoperatively. Then protocol followed for titration of midazolam up to 2 mg IV at beginning and during case.
- Midazolam + Ketamine 5 mg: Drug: Ketamine 10 MG/ML: 0.5 ML
  Ketamine 10 MG/ML: 0.5 ML: 5 mg ketamine IV given just prior to onset of case. Then titrated midazolam up to 2 mg IV at beginning and during case.
- Midazolam + Ketamine 10 mg: Drug: Ketamine 10 MG/ML: 1 ML
  Ketamine 10 MG/ML: 1 ML: 10 mg ketamine IV given just prior to onset of case. Then titrated midazolam up to 2 mg IV at beginning and during case.
Period: Overall Study
Arm/Group | Midazolam Alone | Midazolam + Ketamine 5 mg | Midazolam + Ketamine 10 mg
Started | 41 | 29 | 35
Completed | 41 | 29 | 35
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam Alone | Midazolam + Ketamine 5 mg | Midazolam + Ketamine 10 mg | Total
Number analyzed (Participants) | 41 | 29 | 35 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 7 | 25
  >=65 years | 31 | 21 | 28 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (8.8) | 69.1 (8.1) | 65.6 (9.8) | 68 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 21 | 53
  Male | 22 | 16 | 14 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 29 | 35 | 105

OUTCOME MEASURES:

1. Primary Outcome: Eye Mobility During Surgery (See Link to Study Protocol for Scale)
Description: Scale of mobility of eye during surgery rate 0 (no movement) to 3 (movement enough to stop surgery).
Time Frame: Intraoperative, end of operation reported
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midazolam Alone | Midazolam + Ketamine 5 mg | Midazolam + Ketamine 10 mg
Number analyzed (Participants) | 41 | 29 | 35
units on a scale | 1.39 (0.63) | 1.41 (0.63) | 1.31 (0.63)

2. Secondary Outcome: Measure of Comfort (See Link to Study Protocol for Scale)
Description: Measure of comfort (0-3; 0=very comfortable to 3=extremely uncomfortable
Time Frame: Obtained on the first day after surgery during the subject's routine postoperative check in the Ophthalmology Clinic.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midazolam Alone | Midazolam + Ketamine 5 mg | Midazolam + Ketamine 10 mg
Number analyzed (Participants) | 41 | 29 | 35
units on a scale | 1.29 (0.62) | 1.18 (0.60) | 1.17 (0.59)

3. Secondary Outcome: PACU Length of Stay
Description: This is obtained from the records as time spent in the PACU (Recovery Room) after surgery.
Time Frame: This will occur one time only, in a range of 20 to 30 minutes after the surgery is completed.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Midazolam Alone | Midazolam + Ketamine 5 mg | Midazolam + Ketamine 10 mg
Number analyzed (Participants) | 41 | 29 | 35
Minutes | 19.2 (7.7) | 19.0 (6.5) | 20.1 (10.7)

4. Secondary Outcome: Nausea
Description: Self-reported incidence of nausea. This will be assessed by asking the subjects once (just prior to discharge from the PACU) whether they experienced any nausea while they were in the PACU (Recovery Room) and will be a measurement of the count of participants that experienced nausea during this period
Time Frame: This will occur from time of entry into PACU to time of departure after their surgery. (One time only, in a range of 20 to 30 minutes after surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam Alone | Midazolam + Ketamine 5 mg | Midazolam + Ketamine 10 mg
Number analyzed (Participants) | 41 | 29 | 35
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Midazolam Alone | Midazolam + Ketamine 5 mg | Midazolam + Ketamine 10 mg
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/29 | 0/35
Other Adverse Events (participants affected / at risk) | 0/41 | 0/29 | 0/35

LIMITATIONS AND CAVEATS:
Study may be a bit underpowered for the small differences between groups in measured outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes